CLINICAL TRIAL: NCT04414124
Title: A Randomized, Open Label, Prospective, Parallel Group Study to Assess the Natural History of COVID-19 and Effects of KB109 in Addition to Supportive Self Care (SSC) Compared to SSC Alone on Measures of Health in Non-hospitalized Patients With Mild-Moderate COVID-19
Brief Title: A Clinical Study to Assess the Natural History of COVID-19 and Effects of KB109 and Supportive Self-care in Outpatients With Mild-to-moderate COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K031-120
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-08

CONDITIONS: Mild-to-moderate COVID-19
Keywords: Microbiome; COVID-19; Corona Virus; Corona Virus Disease; Kaleido; Kaleido Biosciences; KB109; Oligosaccharide; Glycan; Pathogens; Microbiome metabolic therapy; MMT; Supportive Self Care; SSC; Telemedicine
MeSH Terms: conditions — COVID-19 | interventions — Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KB109 + Self Supportive Care (SSC) (Other)
  Interventions: Other: KB109 + Self Supportive Care (SSC)
- Self Supportive Care (SSC) Alone (Other)
  Interventions: Other: Self Supportive Care (SSC) Alone

INTERVENTIONS:
Other: KB109 + Self Supportive Care (SSC) — KB109 is a novel glycan
  Arms: KB109 + Self Supportive Care (SSC)
Other: Self Supportive Care (SSC) Alone — Self Supportive Care (SSC) Alone
  Arms: Self Supportive Care (SSC) Alone

SUMMARY:
This randomized, open-label, prospective, parallel-group controlled clinical study that aims to explore the natural history of COVID-19 illness and the safety of KB109, a novel glycan, plus SSC versus SSC alone and measures of health in outpatients with mild-to-moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Be male or female, ≥18 years of age
* Be willing and able to give informed consent
* Screening/Randomization telemedicine visit within 2 days of testing positive test for COVID-19
* Having self-reported fever or cough for not more than 72 hours prior to COVID-19 testing
* Mild to moderate COVID-19
* Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Patients who are hospitalized for in-patient treatment or currently being evaluated for potential hospitalization at the time of informed consent for conditions other than COVID- 19
* History of chronic lung disease
* Ongoing requirement for oxygen therapy
* Shortness of breath in resting position
* Diagnosis of sleep apnea requiring Bilevel Positive Airway Pressure (BIPAP) / Continuous Positive Airway Pressure (CPAP)
* Female patients who are pregnant, trying to become pregnant or lactating
* Is considered, in the opinion of the PI, to be unlikely for any reason to be able to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2020-08-02 (Actual); Primary Completion 2021-02-02 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing study-product related treatment-emergent adverse events (TEAEs) | Day 1 to Day 35

SECONDARY OUTCOMES:
Change from baseline to end of intake in overall composite COVID-19 symptom score | Day 1 to Day 35
  The composite COVID-19 symptom score is the sum of the 8 cardinal COVID-19 related symptom scores (cough, chills/repeated shaking with chills, muscle pain, fever, headache, anosmia/ageusia, shortness of breath, and sore throat). Each COVID-19 symptom will be recorded by patients on a scale of 0: Absent, 1: Mild: Moderately severe. The overall composite score ranges from 0 (no symptoms) to 24 (very severe)
Time to resolution of fever | Day 1 to Day 35
  Resolution of fever is defined as from Day 1 until the day at which a patient's daily maximum temperature achieves and remains below 100.4 Degrees Fahrenheit for the rest of the intake period and for the follow-up period without an antipyretic medication.
Proportion of patients with decreased oxygen saturation | Day 14, Day 35
Effect of COVID-19 symptoms on physical activities | Day 1 to Day 35
  Effect of COVID-19 symptoms on physical activities rated as: not at all, very little, somewhat, quite a lot, could not do physical activities.
Proportion of patients requiring hospitalization | Day 1 to Day 35
Time to resolution of overall 13 COVID-19 related symptoms. | Day 1 to Day 35
  Defined as from Day 1 until the day at which the overall composite score of 13 COVID-19 related symptoms becomes 0 or 1 and remains at 0 or 1 for the rest of the Intake Period and for the Follow-up Period. Overall composite score of 13 COVID-19 related symptoms is the sum of 13 COVID-19 related symptom scores (i.e., cough, chills/repeated shaking with chills, muscle pain, fever, headache, anosmia/ageusia, shortness of breath, sore throat, gastrointestinal disturbance/symptoms, diarrhea, fatigue, nasal congestion, and chest tightness (CDC 2020). Each COVID-19 symptom will be recorded by patients on a scale of 0: Absent, 1: Mild, 2: Moderately severe, 3: Very severe. The overall composite score ranges from 0 (no symptoms) to 39 (very severe).
Time to resolution of overall 8 cardinal COVID-19 related symptoms. | Day 1 to Day 35
  Defined as from Day 1 until the day at which the overall composite score of 8 cardinal COVID-19 related symptoms 0 or 1 and remains at 0 or 1 for the rest of the Intake Period and for the Follow-up Period. Overall composite score of 8 cardinal COVID-19 related symptoms is the sum of 8 cardinal COVID-19 related symptom scores (i.e., cough, chills/repeated shaking with chills, muscle pain, fever, headache, anosmia/ageusia, shortness of breath, and sore throat).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (16):
- United States (16):
  - Healthstar Research, Hot Springs, Arkansas
  - Axon Clinical Research, Riverside, California
  - Medical Center for Clinical Research, San Diego, California
  - Vista Health Research, Miami, Florida
  - Bio-Medical Research, Miami, Florida
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Centex Studies, Inc. - Lake Charles, Lake Charles, Louisiana
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Wake Research - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - Carolina Institute For Clinical Research, Fayetteville, North Carolina
  - M3 Wake Research, Inc, Raleigh, North Carolina
  - TruCare Internal Medicine and Infectious Diseases, DuBois, Pennsylvania
  - ClinSearch LLC, Chattanooga, Tennessee
  - Global Medical Research, DeSoto, Texas
  - Centex Studies, Houston, Texas
  - Infectious Diseases Associates of Central Virginia, Lynchburg, Virginia